CLINICAL TRIAL: NCT06030167
Title: Insecure Attachment and Psychosocial Functioning in Autistic Adults Are Mediated by Depression and Paranoid Ideation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parnassia Groep (Other)
Responsible Party: Principal Investigator, Richard Vuijk, Principal Investigator, Parnassia Groep
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CWO-27-004
Record Dates: First submitted 2023-07-26; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; Attachment; Psychosocial functioning; Adults
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Psychosocial Functioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessment of attachment and psychosocial functioning in adults with ASD (Other): Questionaires about attachment, psychosocial functioning, depressive symptoms, paranoid ideation, and emotion regulation were administered to 83 autistic adults (50 males, 33 females).
  Interventions: Behavioral: Insecure attachment and psychosocial functioning in autistic adults

INTERVENTIONS:
Behavioral: Insecure attachment and psychosocial functioning in autistic adults — Questionaires about attachment, psychosocial functioning, depressive symptoms, paranoid ideation, and emotion regulation were administered to 83 autistic adults (50 males, 33 females).

SUMMARY:
The present study examines if depressive symptoms, paranoid ideation, and emotion regulation strategies mediate the relationship between attachment and psychosocial functioning in autistic adults.

DETAILED DESCRIPTION:
The present study examines if depressive symptoms, paranoid ideation, and emotion regulation strategies mediate the relationship between attachment and psychosocial functioning in autistic adults. Within a cross-sectional design, we used mediation analysis to clarify the roles of co-occurring mental conditions as depressive symptoms, paranoid ideation, and (mal)adaptive emotion regulation strategies in mediating the pathway from insecure attachment to psychosocial functioning in autistic adults. Questionaires about attachment, psychosocial functioning, depressive symptoms, paranoid ideation, and emotion regulation were administered to 83 autistic adults (50 males, 33 females).

ELIGIBILITY:
Inclusion Criteria:

* a primary clinical diagnosis of DSM-5 ASD (APA, 2013)
* age ≥ 18 years
* at least eight years of education.

Exclusion Criteria:

* intellectual disability (IQ ≤ 80)
* presence of current suicidal ideation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Experiences in Close Relationships - Revised questionnaire (ECR-r) | 15 minutes
  Measuring self-rated levels of insecure attachment in 83 adults with autism spectrum disorder. Welch's two sample t-test was used to compare the ECR-r data between the participants and (non-)clinical controls drawn from the manuals of the used measure.
  The ECR-R is a 36-item measure designed to assess individual differences with respect to attachment-related anxiety (i.e., the extent to which people are insecure versus secure about the availability and responsiveness of romantic partners; items 1 to 18) and attachment-related avoidance (i.e., the extent to which people are uncomfortable being close to others versus secure depending on others; items 19 to 36). The items are scored on a 7-point scale, with higher scores (>= 4) indicating more insecure attachment. A mean score (ranging from 0 to 7) is calculated for both attachment styles.
World Health Organisation Disability Assessment Schedule 2.0 (WHODAS 2.0) | 15 minutes
  Measuring self-rated levels of psycho-social functioning in 83 autistic adults. Welch's two sample t-test was used to compare the WHODAS 2.0 data between the participants and (non-)clinical controls drawn from the manuals of the used measure.
  WHODAS 2.0 is a generic assessment self-report for health and disability in adults, consisting of 36 items on a 5-point scale (none, mild, moderate, severe, and extreme) covering six domains: cognitions, mobility, self-care, interaction, life activities, and participation in society. WHODAS 2.0 asks the individual to rate how much difficulty they have had in specific areas of functioning during the past 30 days. WHODAS 2.0 produces standardized disability levels and profiles by summing six domain scores and converting the summary score into a metric range from 0 (= no disability) to 100 (= full disability).

SECONDARY OUTCOMES:
Beck Depression Inventory-Second Edition-Dutch version-Revised (BDI-2-NL-R) | 10 minutes
  Measuring self-rated levels of depression in 83 autistic adults. Welch's two sample t-test was used to compare the BDI-2-NL-R data between the participants and (non-)clinical controls drawn from the manuals of the used measure.
  The BDI-2-NL-R is a 21-item self report assessing the presence and severity of depressive symptoms, according to the Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition (DSM-IV; American Psychiatric Association, 1994). The BDI-2-NL-R is also compatible with DSM-5 depressive disorder (APA, 2013; 2022). The items are scored on a 4-point scale with a total score ranging from 0 to 63 indicating minimal (0-13), mild (14-19), moderate (20-28), or severe (29-63) depression.
Green Paranoid Thought Scales (GPTS) | 15 minutes
  Measuring self-rated levels of paranodi thoughts in 83 autistic adults. Welch's two sample t-test was used to compare the GPTS data between the participants and (non-)clinical controls drawn from the manuals of the used measure.
  The GPTS is a 32-item self-report assessing 16 ideas of persecution and 16 ideas of social reference on a 5-point scale, with a total score ranging from 32 to 160, with higher scores indicating higher levels of paranoid ideation.
FEEL-E Questionnaire for Emotion Regulation in Adults (FEEL-E) | 20 minutes
  Measuring self-rated levels of emotion regulation in 83 autistic adults. Welch's two sample t-test was used to compare the GPTS data between the participants and (non-)clinical controls drawn from the manuals of the used measure.
  The FEEL-E is a 72-item self-report questionnaire assessing emotion regulation strategies, consisting of six adaptive (problem-oriented action, acceptance, cognitive problem-solving, reappraisal, evoking positive feelings, forgetting) and six maladaptive (withdrawal, self-blame, resignation, rumination, negative thinking, other-blame) strategies. The items are scored on a 5-point scale with a total score ranging from 36 to 180 for each strategy (T-score < 40: below average use of strategy; T-score 40-60: average use of strategy; T-score > 60: above average use of strategy).

CONTACTS AND LOCATIONS:
Overall Officials: Richard Vuijk, Dr., Principal Investigator — Parnassia Antes
Locations (1):
- Parnassia Antes, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No